CLINICAL TRIAL: NCT04517110
Title: Peri-Operative Pregabalin for Reducing opIoid Consumption AfTer Cardiac surgEry: A Randomized Trial
Brief Title: Perioperative Pregabalin for Reducing Opioid Consumption After Cardiac Surgery
Acronym: OPIATE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The COVID-19 pandemic has reduced recruitment such that the study is no longer feasible
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Andre Lamy, Cardiac Surgeon, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPIATE-2020
Record Dates: First submitted 2020-08-11; First posted 2020-08-18 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Opioid Use
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebo capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pregabalin + Usual Care (Experimental): 300 mg pregabalin taken orally within 2 hours before surgery and 75 mg pregabalin taken orally twice daily after surgery beginning after successful extubation (day after surgery or later) until discharge or 5 days, whichever comes first. Participants will also receive standard pain management.
  Interventions: Drug: Pregabalin 300 mg; Drug: Pregabalin 75 mg; Other: Usual Care
- Placebo + Usual Care (Placebo Comparator): Placebo taken orally within 2 hours before surgery and placebo taken orally twice daily after surgery beginning after successful extubation (day after surgery or later) until discharge or 5 days, whichever comes first. Participants will also receive standard pain management.
  Interventions: Drug: Pregabalin 300 mg Placebo; Drug: Pregabalin 75 mg Placebo; Other: Usual Care

INTERVENTIONS:
Drug: Pregabalin 300 mg — Pregabalin 300 mg, capsule
  Other Names: Lyrica
  Arms: Pregabalin + Usual Care
Drug: Pregabalin 75 mg — Pregabalin 75 mg twice daily, capsules
  Other Names: Lyrica
  Arms: Pregabalin + Usual Care
Drug: Pregabalin 300 mg Placebo — Placebo, matching Pregabalin 300 mg capsule
  Other Names: Placebo Capsule
  Arms: Placebo + Usual Care
Drug: Pregabalin 75 mg Placebo — Placebo, matching Pregabalin 75 mg capsules
  Other Names: Placebo Capsule
  Arms: Placebo + Usual Care
Other: Usual Care — Usual Care

SUMMARY:
OPIATE is a double-blinded randomized controlled trial (RCT) comparing pregabalin in addition to usual care to usual care alone for reducing post-operative opioid consumption in patients undergoing on-pump cardiac surgery. Patients will be randomized in a 1:1 ratio to receive either pregabalin (300 mg pre-operatively + 75 mg post-operatively twice daily until discharge or 5 days) in addition to usual care or matching placebos in addition to usual care. The aim of the trial is to show that pregabalin is superior to usual care (i.e. a superiority trial).

DETAILED DESCRIPTION:
By administering oral pregabalin to patients before and after cardiac surgery for pain relief, we aim to reduce the amount of opioids they will require for pain relief and reduce opioid-related side effects that they may experience after surgery. Participants will be randomly assigned to receive either pregabalin in addition to usual care or usual care alone. Participants in the pregabalin group will receive two 150 mg pregabalin capsules (300 mg total dose) within 2 hours before surgery and a 75 mg pregabalin capsule twice daily after surgery until discharge from hospital to a maximum of 5 days after surgery. Participants in the usual care group will receive two placebo study capsules within 2 hours before surgery and a placebo capsule twice daily after surgery until discharged from hospital to a maximum of 5 days after surgery. OPIATE will be the largest clinical trial of pregabalin in cardiac surgery with results that are expected to set new post-operative pain management guidelines to encourage the widespread use of pregabalin in cardiac patients.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Undergoing cardiac surgery with median sternotomy
3. Provide written informed consent

Exclusion Criteria:

1. Use of opioids or cannabis products in the past 30 days
2. Daily use of pregabalin or gabapentin within 7 days of randomization
3. Intravenous drug user
4. Have a hypersensitivity or allergy to pregabalin
5. History of previous cardiac surgery
6. Undergoing minimally invasive surgery
7. Emergency surgery
8. Severe renal impairment (creatinine > 250 μmol/L)
9. Unable to swallow study medications
10. Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Cumulative opioid consumption | After surgery until discharge from hospital or 5 days, whichever is first.
  Dose of opioids consumed (in morphine equivalents) by participants
Daily opioid consumption | Each postoperative day, beginning on postoperative day 1 and ending on the day of discharge from hospital or postoperative day 5, whichever is first.
  Dose of opioids consumed (in morphine equivalents) by participants

SECONDARY OUTCOMES:
Daily postoperative pain | Each postoperative day, beginning on postoperative day 1 and ending on the day of discharge from hospital or postoperative day 5, whichever is first.
  Acute postoperative pain assessed by the numeric rating scale (NRS; 0 to 10)
Average postoperative pain | Average of scores after surgery until discharge from hospital or 5 days, whichever is first.
  Acute postoperative pain assessed by the numeric rating scale (NRS; 0 to 10)
Cumulative consumption of antiemetic medications | After surgery until discharge from hospital or 5 days, whichever is first.
  Dose of gravol or ondansetron consumed by participants
Daily consumption of antiemetic medications | Each postoperative day, beginning on postoperative day 1 and ending on the day of discharge from hospital or postoperative day 5, whichever is first.
  Dose of gravol or ondansetron consumed by participants
Time to extubation | Within the first 5 days after surgery
  Time from surgery completion until first successful extubation
Mobility | Within the first 5 days after surgery
  Proportion of mobility goals met after surgery
Delirium | Starting the second day after surgery and ending after 5 days or 3 days of negative tests.
  Number of participants meeting the Confusion Assessment Method (CAM) criteria
Major adverse cardiovascular events | Within the first 5 days after surgery
  The first occurrence of death, non-fatal myocardial infarction (MI) or non-fatal stroke
Death | Within the first 5 days after surgery
  Number of participants experiencing death from any cause
Myocardial infarction | Within the first 5 days after surgery
  Number of participants experiencing myocardial infarction (MI) without death
Stroke | Within the first 5 days after surgery
  Number of participants experiencing stroke without death

CONTACTS AND LOCATIONS:
Overall Officials: Andre Lamy, MD, MHSc, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pesonen A, Suojaranta-Ylinen R, Hammaren E, Kontinen VK, Raivio P, Tarkkila P, Rosenberg PH. Pregabalin has an opioid-sparing effect in elderly patients after cardiac surgery: a randomized placebo-controlled trial. Br J Anaesth. 2011 Jun;106(6):873-81. doi: 10.1093/bja/aer083. Epub 2011 Apr 6. PMID 21474474
- [Background] Joshi SS, Jagadeesh AM. Efficacy of perioperative pregabalin in acute and chronic post-operative pain after off-pump coronary artery bypass surgery: a randomized, double-blind placebo controlled trial. Ann Card Anaesth. 2013 Jul-Sep;16(3):180-5. doi: 10.4103/0971-9784.114239. PMID 23816671
- [Background] Sundar AS, Kodali R, Sulaiman S, Ravullapalli H, Karthekeyan R, Vakamudi M. The effects of preemptive pregabalin on attenuation of stress response to endotracheal intubation and opioid-sparing effect in patients undergoing off-pump coronary artery bypass grafting. Ann Card Anaesth. 2012 Jan-Mar;15(1):18-25. doi: 10.4103/0971-9784.91473. PMID 22234017
- [Background] Ziyaeifard M, Mehrabanian MJ, Faritus SZ, Khazaei Koohpar M, Ferasatkish R, Hosseinnejad H, Mehrabanian M. Premedication with oral pregabalin for the prevention of acute postsurgical pain in coronary artery bypass surgery. Anesth Pain Med. 2015 Jan 17;5(1):e24837. doi: 10.5812/aapm.24837. eCollection 2015 Feb. PMID 25830118
- [Background] Bouzia A, Tassoudis V, Karanikolas M, Vretzakis G, Petsiti A, Tsilimingas N, Arnaoutoglou E. Pregabalin Effect on Acute and Chronic Pain after Cardiac Surgery. Anesthesiol Res Pract. 2017;2017:2753962. doi: 10.1155/2017/2753962. Epub 2017 Apr 30. PMID 28539936
- [Background] Anwar S, Cooper J, Rahman J, Sharma C, Langford R. Prolonged Perioperative Use of Pregabalin and Ketamine to Prevent Persistent Pain after Cardiac Surgery. Anesthesiology. 2019 Jul;131(1):119-131. doi: 10.1097/ALN.0000000000002751. PMID 31149930